CLINICAL TRIAL: NCT06052410
Title: The Effect of Early Intervention on Sensory, Cognitive and Motor Outcomes in Children at Risk of Developmental Delay: A Randomized Controlled Study
Brief Title: Early Intervention in Children at Risk of Developmental Delay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ezginur Gündoğmuş, Occupational Therapist, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Hacettepe Occupational Therapy
Record Dates: First submitted 2023-09-19; First posted 2023-09-25 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Developmental Delay
Keywords: early intervention; developmental delay; motor development; cognitive development
MeSH Terms: conditions — Learning Disabilities | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: Sensory development is targeted in activity-based education based on the principles of the Goal, Activity and Motor Enrichment (GAME) approach, which is an evidence-based early intervention approach for children between 24-36 months at risk of developmental delay. The program was implemented in the pediatric unit for 45 minutes a day, twice a week for 12 weeks. For the control group, evaluation tests were first applied to babies selected by simple random sampling method. According to the evaluation results, a personalized home program was given. Post-evaluations were repeated for both groups after 12 weeks. The basic principles of the GAME approach are examined in 3 parts: goal-oriented intensive motor training, parent training, environmental enrichment. In our study, activities were also implemented based on the sensory integration approach and cognitive rehabilitation intervention principles to present sensory and cognitive strategies within the activity.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Other): The group in which the early intervention program was implemented.
  Interventions: Other: Early Intervention
- Control Group (Other): The group where the home program is applied
  Interventions: Other: Home Programme

INTERVENTIONS:
Other: Early Intervention — Based on the principles of the Goal, Activity and Motor Enrichment (GAME) approach, which is an evidence-based early intervention approach for children at risk of developmental delay between 24-36 months, activity-based training is aimed at the development of sensory and cognitive skills in addition to the training of motor skills, which are intensively discussed in the content of the approach. Individualized early occupational therapy intervention including strategies was implemented.
  Arms: Intervention Group
Other: Home Programme — For the control group, evaluation tests were first applied to the babies selected by simple random sampling method. An individualized home program was given according to the evaluation results. Home programs include activities for every skill area and were prepared together with the parents, taking into account the criteria suggested for the success of the home program. Based on these criteria, it was checked whether the family had received another home program, and while preparing the program, care was taken not to overload the parents, importance was given to the family's willingness to receive the home program, activities and goals were decided in cooperation with the parent, thus facilitating the applicability of the activities in daily life, ensuring that the number of activities was 6. Care was taken to ensure that the activity was not too much, the parent was given the necessary time to implement the program, and a phone call was made to the parent every 3 weeks.
  Arms: Control Group

SUMMARY:
Although it is stated in the literature that development should be considered as a whole and sensory, cognitive and motor outcomes are interrelated, it is seen that interventions for sensory and cognitive skills are not included in early intervention studies. For this reason, the study examined the effects of an early occupational therapy intervention program, which includes sensory, cognitive and motor strategies based on the principles of Goal, Activity and Motor Enrichment-GAME, an evidence-based early intervention program, on the sensory, cognitive and motor skills of babies at risk of developmental delay for 24-36 months.

DETAILED DESCRIPTION:
Children with developmental delays benefit from early intervention. Therefore, it is very important to detect developmental delays as early as possible. In recent years, there has been increasing interest in designing and providing early intervention programs to improve developmental outcomes for infants at risk for developmental delay for neurodevelopmental disorders. Early intervention includes services provided to children from birth to age five to promote the child's health and well-being, develop emerging skills, minimize developmental delays, correct existing or emerging disabilities, prevent functional impairment, and promote parental compliance. When the literature is examined, it is seen that early intervention approaches are mostly implemented in preterm babies and focus on motor skills. An example of studies carried out with this attitude is Neurodevelopmental Treatment (NGT), which is frequently used in early intervention approaches in Turkey. Another early intervention approach that includes intensive motor training is Goal, Activity and Motor Enrichment (GAME). GAME early intervention approach is also used in extremely preterm babies with a high risk of developmental delay; It has been used in studies as an intervention approach that includes goal-oriented motor training, environmental enrichment and family education. Another early intervention approach that addresses parent education and environmental enrichment principles is the Supporting Play, Exploration and Early Development Intervention (SPEEDI). The SPEEDI program was applied to preterm babies in a similar way to the GAME program. Other approaches used by occupational therapists for children at risk of developmental delay in the literature are home-based and routine-based approaches.

When the literature is examined, it is seen that early intervention programs are mostly carried out with premature babies and/or for the diagnosis of cerebral palsy (CP). Early intervention approaches in the literature include intensive motor training, parent training, environmental enrichment, participation support and home visits. Although it is stated in the literature that development should be considered as a whole and sensory, cognitive and motor outcomes are interrelated, it is seen that interventions for sensory and cognitive skills are not included in early intervention studies. Therefore, the aim of our study is to improve the sensory, cognitive and motor skills of the early occupational therapy intervention program, which includes sensory, cognitive and motor strategies based on the principles of Goal, Activity and Motor Enrichment-GAME, which is an evidence-based early intervention program, in babies at risk of developmental delay of 24-36 months. to examine its effect.

ELIGIBILITY:
Inclusion Criteria:

1. Being at risk of developmental delay between 24 and 36 months
2. Not having received any neurological, psychiatric or orthopedic diagnosis,
3. The family is willing to participate in the study and agrees to participate regularly in the intervention program and evaluations.

Exclusion Criteria:

1. Babies staying in institutional care,
2. Having any neurological, psychiatric or orthopedic diagnosis

Ages: 24 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2022-09-03 (Actual); Primary Completion 2022-11-26 (Actual); Study Completion 2022-12-03 (Actual)

PRIMARY OUTCOMES:
Infants/Toddler Sensory Profile 2 (ITSP 2) | 10 minutes
  It is a 5-point Likert type scale filled out by families that evaluates the sensory processing skills of children aged 7-35 months.

SECONDARY OUTCOMES:
Bayley Scales of Infant and Toddler Development III (Bayley III), | 40 minutes
  It is a scale in which children's gross motor, fine motor, communication and cognitive skills are evaluated by the therapist.
Ages and Stages Questionnaire (ASQ) and Ages and Stages Questionnaire- Social Emotional (ASQ-SE). | 45 minutes
  It is a scale in which children's gross motor, fine motor, communication, cognitive and social emotional skills are evaluated by the family.

CONTACTS AND LOCATIONS:
Overall Officials: Ezginur Gündoğmuş, Study Director — OT MSc
Locations (1):
- Hacettepe University, Ankara, Altındag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Participants' data are stored with the researcher by giving them a code. It is not planned to be shared with any person or institution.